CLINICAL TRIAL: NCT06360614
Title: The Effect of Hand Massage Applied to Palliative Care Oncology Patients on Pain, Comfort and Sleep Quality
Brief Title: The Effect of Hand Massage Applied to Palliative Care Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: murat koç (Other Government)
Collaborators: Istanbul Sultanbeyli State Hospital (Other Government)
Responsible Party: Sponsor-Investigator, murat koç, Investigator, Istanbul Sultanbeyli State Hospital
Organization: Istanbul Sultanbeyli State Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2024s01
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Hand Massage
Keywords: Palliative care; Oncology; Hand massage; Pain; Comfort; Sleep quality
MeSH Terms: conditions — Neoplasms; Pain; Sleep Initiation and Maintenance Disorders | interventions — Nursing Care

STUDY DESIGN:
Intervention Model Description: Before the application, data will be collected and recorded through a face-to-face interview (8-10 minutes) by a nurse who does not know which group the patients are in. Sleep times of patients will be measured with a smart bracelet. At this stage, the same procedure will be continued for the intervention and control groups.
  Hand massage will be applied to the intervention group for 4 weeks, 2 days a week (Monday and Friday), 2 sessions each day. The control group will receive routine monitoring and nursing care for 4 weeks.
  In the intervention and control groups, VAS-Pain, General Comfort Scale and Pittsburgh Sleep Quality were assessed by a face-to-face interview by a nurse who did not know which group the patients were in, on the 7th day (Monday), 14th day (Monday) and 28th day (Monday). Index measurement tools will be applied and patients' sleep times will be measured with a smart bracelet.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hand massage application (Experimental): Hand massage will be applied to the intervention group for 4 weeks, 2 days a week (Monday and Friday), 2 sessions each day.
  Interventions: Other: Hand massage application
- Control Group (Placebo Comparator): The control group will receive routine monitoring and nursing care for 4 weeks.
  Interventions: Other: routine monitoring and nursing care

INTERVENTIONS:
Other: Hand massage application — 2 sessions of hand massage every day, 2 days a week (Monday and Friday) for 4 weeks
  Arms: Hand massage application
Other: routine monitoring and nursing care — Routine monitoring and nursing care for 4 weeks
  Arms: Control Group

SUMMARY:
World Health Organization (WHO) palliative care is defined as "an approach that aims to reduce or prevent suffering by early identification, evaluation and treatment of the physical, psychosocial and spiritual problems of patients and families accompanying life-threatening diseases, and thus to increase their quality of life." Palliative care is a multidisciplinary approach that provides appropriate health care for oncology patients, who have a wide variety of medical, functional, social and emotional needs. Pharmacological approaches are generally used in symptom management of palliative care patients. In addition to pharmacological approaches, non-pharmacological approaches are also preferred. Massage is a preferred intervention among professional nursing practices because it is reliable, has no side effects, has a direct effect on patients, and is easy to apply.

Massage is the stimulation of the skin, subcutaneous tissue, muscles, internal organs, metabolism, circulation and lymph systems for therapeutic purposes through mechanical and neural means. The presence of sufficient mechanoreceptors in the hands, which stimulate painless nerve endings, shows that the hands should be chosen as the appropriate area for massage. Among the effects of hand massage: ensuring the regeneration of cells, facilitating the elimination of accumulated toxins, providing relaxation, helping to reduce pain by facilitating the release of endorphins, helping to increase circulation, regulating respiratory functions, providing stress and anxiety control, creating a state of well-being, strengthening the immune system, increasing general comfort, improving sleep quality. is located. Studies in the literature have found that hand massage reduces anxiety levels, stress and agitation levels, pain levels, and increases comfort and sleep levels. As seen in the literature, the effectiveness of hand massage applied to different sample groups on anxiety, stress, agitation, pain, comfort and sleep parameters was evaluated. There are very few studies evaluating the effectiveness of hand massage applied to oncology patients. In addition, no study has been found that evaluated the effects of hand massage on pain, comfort and sleep in palliative oncology patients, who constitute the majority of palliative care patients.

DETAILED DESCRIPTION:
There is a rapid increase in cancer incidence and mortality worldwide. The International Agency for Research on Cancer (IARC) 2018 found that 18.1 million individuals were diagnosed with cancer worldwide. Individuals diagnosed with cancer experience many symptoms during the disease process, during the treatment phase, and in the terminal period. In most patients, many symptoms such as pain, insomnia, nausea and vomiting, anorexia, shortness of breath and fatigue are frequently observed, depending on the type and stage of cancer, treatments applied and accompanying diseases. Failure to control these symptoms affects the treatment process and may cause patients and family members to experience difficulties in the fight against cancer. During this period, the most effective way to meet all the needs of the patient and his family is to receive palliative care services. Palliative care is the key to individualized and holistic care. The scope of palliative care includes defining goals of care based on the patient's values and beliefs and addressing patients' physical, emotional, spiritual, and social problems. Palliative care is a multidisciplinary approach in which appropriate health care is provided for oncology patients, who have a wide range of medical, functional, social and emotional needs. Pharmacological approaches are generally used in symptom management of palliative care patients. In addition to pharmacological approaches, non-pharmacological approaches are also preferred. Practices such as reflexology, music therapy, acupuncture, aromatherapy, pet therapy, therapeutic touch, reiki, massage, hand massage therapy are non-pharmacological applications that can be used in palliative care oncology patients.

Massage is a preferred intervention among professional nursing practices because it is reliable, has no side effects, has a direct effect on patients, and is easy to apply. Massage is the stimulation of the skin, subcutaneous tissue, muscles, internal organs, metabolism, circulation and lymph systems for therapeutic purposes through mechanical and neural means . The presence of sufficient mechanoreceptors in the hands, which stimulate painless nerve endings, shows that the hands should be chosen as the appropriate area for massage. Hand massage application changes the sensation of pain in the neuromatrix. It increases the stimulation of large nerve fibers on the small C nerve fiber in the spinothalamic system through the spinal cord and reduces the sensation and transmission of pain by increasing blood flow to the hands. With the application of hand massage, sensory information is transferred from the hands to the spinothalamic pathway via the thalamus and somatosensory cortex via the spinal cord. While sensory information changes within the neuromatrix structure, it also reduces chronic pain. The scope of hand massage is limited, but it is a more accessible area. In addition, it can be applied more easily and conveniently than whole body massage due to its pain-reducing and comfort-increasing effect Among the effects of hand massage: ensuring the regeneration of cells, facilitating the elimination of accumulated toxins, providing relaxation, helping to reduce pain by facilitating the release of endorphins, helping to increase circulation, regulating respiratory functions, providing stress and anxiety control, creating a state of well-being, strengthening the immune system, increasing general comfort, improving sleep quality. Studies in the literature show that hand massage reduces anxiety levels, pain levels, stress and agitation levels; It has been stated that it is effective in increasing the level of comfort and sleep quality.

As seen in the literature, the effectiveness of hand massage applied to different sample groups on anxiety, stress, agitation, pain, comfort and sleep parameters was evaluated. There are very few studies evaluating the effectiveness of hand massage applied to oncology patients. In addition, no study has been found that evaluated the effects of hand massage on pain, comfort and sleep in palliative oncology patients, who constitute the majority of palliative care patients. Hand massage, which is a practical, safe and cost-free method in symptom management, which forms the basis of palliative care and has an important place in the treatment of oncology patients, should be used by evaluating its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Oncology patients receiving treatment for at least 2 weeks in palliative care.
* 18 years and over.
* Able to communicate clearly and effectively.
* Visual Analogue Scale-Pain score above 3.
* Pittsburgh Sleep Quality Index score above 5.
* Without a neurological medical diagnosis.
* There is no intravenous catheter on the hand and there is no deformity in the hand.

Exclusion Criteria:

* Less than 2 weeks of treatment in palliative care.
* Under 18 years of age.
* Outside the clinical protocol use analgesic medication or methods.
* A change in the standard protocol for pain and sleep.
* Visual Analogue Scale-Pain score below 3.
* Pittsburgh Sleep Quality Index score below 5.
* Unable to communicate effectively.
* Patients with diagnosed neurological problems and hand deformities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-19 (Actual)

PRIMARY OUTCOMES:
İndividual Information Form | 4 weeks
  Prepared by the researcher in accordance with the purpose of the research. The Personal Information Form consists of questions about individuals' socio-demographic characteristics, pain and sleep patterns.
Patient Follow-up Form | 4 weeks
  It was prepared by the researcher in accordance with the purpose of the study. The Patient Monitoring Form allows recording of VAS-Pain, General Comfort Scale and Pittsburgh Sleep Quality Index scores evaluated on days 0, 7, 14 and 28.
General Comfort Scale | 4 weeks
  It is used to determine the needs in providing comfort and to evaluate the results of nursing interventions aimed at comfort. The General Comfort Scale, which is suitable for Turkish society by Kuğuoğlu and Karabacak (2004), is a four- and six-point Likert type, contains 24 positive and 24 negative items, and the response patterns are mixed.
  The highest total score to be obtained from the scale is 192, and the lowest total score is 48. The average value is determined by dividing the total score obtained by the number of scale items and the result is stated as 20 in the 1-4 distribution. Thus, the comfort level; Low comfort is expressed in a range of one point and high comfort is expressed in a range of four points. As a result of the Turkish validity-reliability study of GKS, it was found that the reliability of the scale was high (Cronbach's alpha = 0.85).
Pittsburgh Sleep Quality Index | 4 weeks
  The validity and reliability study of the scale in our country (Cronbach Alpha = 0.80) was conducted by Ağargün et al. in 1996. PSQI, which evaluates sleep quality in the last month, contains a total of 24 questions. 19 of these are self-report questions and are answered by the patient, while 5 questions are answered by a spouse or a roommate and are used only for clinical information and are not included in scoring. The scale consists of seven components: Subjective Sleep Quality, Sleep Latency, Sleep Duration, Sleep Efficiency, Sleep Disorder, Sleeping Medication Use, and Daytime Dysfunction. In the scale scoring, Subjective Sleep Quality, Sleep Duration and Sleeping Medication Use components are scored between 0-3 depending on the answer given. The total score obtained varies between 0-21 points, and high scores indicate poor sleep quality and high level of sleep disturbance. A total score of 5 or more from the scale indicates that sleep quality is significantly poor.
Smart Bracelet | 4 weeks
  Recording sleep/wake data of patients receiving hand massage; Smart bracelets were used to monitor sleep quality and process. The smart bracelet tracks your sleep patterns and provides information such as the time you fell asleep, the time you woke up, how many times you woke up during the night, and how long it took you to fall asleep each time. The sleep time measured by the smart bracelet is accessed through applications installed on smartphones by the researcher. Xiaomi Smart band 8 Pro was used to measure sleep times. The calibration of the device was carried out monthly at Xiaomi authorized service.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Koç, Principal Investigator — Istanbul Sultanbeyli State Hospital; Nurdan Yalçın ATAR, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Sultanbeyli State Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris D. Safe and effective prescribing for symptom management in palliative care. Br J Hosp Med (Lond). 2019 Dec 2;80(12):C184-C189. doi: 10.12968/hmed.2019.80.12.C184. PMID 31822173
- [Background] Hokka M, Kaakinen P, Polkki T. A systematic review: non-pharmacological interventions in treating pain in patients with advanced cancer. J Adv Nurs. 2014 Sep;70(9):1954-1969. doi: 10.1111/jan.12424. Epub 2014 Apr 15. PMID 24730753
- [Background] Askan F, Lafci Bakar D. The Effect of Hand Massage on Preoperative Anxiety Level and Hemodynamic Variables in Children: A Randomized Controlled Trial. J Perianesth Nurs. 2023 Oct;38(5):773-781. doi: 10.1016/j.jopan.2023.01.013. Epub 2023 Jul 15. PMID 37452817
- [Background] Demir B, Saritas S. Effect of hand massage on pain and anxiety in patients after liver transplantation: A randomised controlled trial. Complement Ther Clin Pract. 2020 May;39:101152. doi: 10.1016/j.ctcp.2020.101152. Epub 2020 Mar 21. PMID 32379634
- [Background] Cavdar AU, Yilmaz E, Baydur H. The Effect of Hand Massage Before Cataract Surgery on Patient Anxiety and Comfort: A Randomized Controlled Study. J Perianesth Nurs. 2020 Feb;35(1):54-59. doi: 10.1016/j.jopan.2019.06.012. Epub 2019 Sep 21. PMID 31551136
- [Background] Schaub C, Von Gunten A, Morin D, Wild P, Gomez P, Popp J. The Effects of Hand Massage on Stress and Agitation Among People with Dementia in a Hospital Setting: A Pilot Study. Appl Psychophysiol Biofeedback. 2018 Dec;43(4):319-332. doi: 10.1007/s10484-018-9416-2. PMID 30209712
- [Background] Gensic ME, Smith BR, LaBarbera DM. The effects of effleurage hand massage on anxiety and pain in patients undergoing chemotherapy. JAAPA. 2017 Feb;30(2):36-38. doi: 10.1097/01.JAA.0000510988.21909.2e. PMID 28098671
- [Background] Cino K. Aromatherapy hand massage for older adults with chronic pain living in long-term care. J Holist Nurs. 2014 Dec;32(4):304-13; quiz 314-5. doi: 10.1177/0898010114528378. Epub 2014 Apr 14. PMID 24733781
- [Background] Kudo Y, Sasaki M. Effect of a hand massage with a warm hand bath on sleep and relaxation in elderly women with disturbance of sleep: A crossover trial. Jpn J Nurs Sci. 2020 Jul;17(3):e12327. doi: 10.1111/jjns.12327. Epub 2020 Feb 3. PMID 32017413
- [Background] Yucel SC, Arslan GG, Bagci H. Effects of Hand Massage and Therapeutic Touch on Comfort and Anxiety Living in a Nursing Home in Turkey: A Randomized Controlled Trial. J Relig Health. 2020 Feb;59(1):351-364. doi: 10.1007/s10943-019-00813-x. PMID 30982141